CLINICAL TRIAL: NCT00299780
Title: Phase I Study of Parathyroid Hormone in Combination With G-CSF in Patients Requiring Additional Stem Cell Mobilization
Brief Title: Safety Study of Parathyroid Hormone in Patients Needing Additional Stem Cell Mobilization.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-109
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Lymphoma; Multiple Myeloma; Acute Myelogenous Leukemia
Keywords: Mobilization; Stem Cell; Parathyroid Hormone
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Leukemia, Myeloid, Acute | interventions — Hematopoietic Stem Cell Mobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Stem cell mobilization

SUMMARY:
The purpose of this study is to determine the safety of parathyroid hormone in combination with G-CSF when used as a stem cell mobilization regimen for patients who fail to mobilize sufficient progenitor stem cells after one or two attempts.

DETAILED DESCRIPTION:
Patients will start treatment within 21 days of the determination of inadequate mobilization. PTH treatment will be given in 4 cohorts: 40 mcg, 60 mcg, 80 mcg, and 10 mcg. PTH will be given on day 1 and continue until stem cell collections are complete or a maximum of 20 days. G-CSF 10 mcg/kg will be given on days 10-14 and continue until stem cell collections are complete. Patients with inadequate CD34+ cells on Day 14 will meet off study criteria and not continue with PTH/G-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Disease status: NHL or HD refractory to chemotherapy, relapsed, o high risk first remission; multiple myeloma; AML in second or subsequent remission or in first remission with adverse cytogenetics or antecedent hematologic disorder.
* Failed one or two mobilization attempts.
* ECOG performance status of 0, 1, or 2.

Exclusion Criteria:

* Cardiac disease: symptomatic congestive heart failure, angina pectoris or uncontrolled hypertension
* Pulmonary disease: severe chronic obstructive lung disease, or symptomatic restrictive lung disease.
* Renal disease: serum creatinine > 2 mg/dl
* Hepatic disease: SGOT or SGPT > 3x normal; serum bilirubin > 2.0 mg/dl that is not due to Gilbert's syndrome or hemolysis
* Calcium > 10.5
* Phosphate < 1.6
* Uncontrolled infection
* Pregnancy or breast feeding mother

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2004-07; Study Completion 2007-04

PRIMARY OUTCOMES:
To assess safety of parathyroid hormone in combination with G-CSF when used as a mobilization agent at four different dosing levels.

SECONDARY OUTCOMES:
To evaluate the peripheral blood CD34+ count after second mobilization.
To evaluate CD34+ cells/kg from apheresis after second mobilization.
To evaluate the percent of patients for whom adequate numbers of CD34+ cells are obtained.
To evaluate transfusion support.
To evaluate the days to neutrophil engraftment (ANC >500) post autologous transplant.
To evaluate the days to platelet engraftment (platelet count > 20,000 unsupported).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ballen, M.D., Principal Investigator — Massachusetts General Hospital, Harvard University
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas